CLINICAL TRIAL: NCT06412029
Title: Understanding and Enhancing Health-Related Social Needs (HRSN) Screening Among Community Oncology Practices
Acronym: HRSN
Status: Enrolling by invitation | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00113288; NCI-2024-02411 (Other: NCI Trial Identifier); WF-2303CD (Other: Lead Organization Identifier); 5UG1CA189824 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-14 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: Cancer Health Disparities
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1: Part 1: Participants attend training, complete clinic assessments and observations and may complete an interview on study.
  Interventions: Other: Non-Interventional
- Part 2: Part 2: Identified clinic staff will be interviewed to discuss factors that influence health related social needs (HRSN) screening at their clinic and help develop generalized guidance.
  Interventions: Other: Non-Interventional
- Part 3: Part 3: Participants attend a co-design workshop and complete surveys on study feasibility.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-interventional study

SUMMARY:
This study evaluates health related social needs screening processes in community oncology clinics.

DETAILED DESCRIPTION:
The primary objective of this study is to assess current processes around health related social needs (HRSN) screening among NCORP clinics and categorize clinics based on their implementation of HRSN screening. The primary endpoint will be a detailed understanding of current processes, with attention to variability by key clinic characteristics.

There are 3 parts of the study in which participants can participate in one or all parts (3 total).

Part 1: Participants attend training, complete clinic assessments and observations and may complete an interview on study.

Part 2: Identified clinic staff will be interviewed to discuss factors that influence HRSN screening at their clinic and help develop generalized guidance.

Part 3: Participants attend a co-design workshop and complete surveys on study feasibility.

ELIGIBILITY:
Inclusion Criteria:

Part 1

NCORP PRACTICES:

* Must be an affiliate or sub-affiliate of an NCORP Community or Minority Underserved Community site
* Must provide outpatient oncology care
* Must be a NCORP practice (defined as one or more NCORP affiliates/sub-affiliates, that have a common administrative structure and share providers and/or patients)
* Must have identified two or more Practice Staff that are available and willing to participate on the Practice Interest Form
* Must have identified at least 1-3 outpatient oncology clinics willing to participate on the Practice Interest Form

CLINICS:

* 1-3 clinics within the practice should be selected
* Clinics may or may not be located in different physical locations
* The investigators will encourage NCORP practices to select clinics within a practice that differ in current or potential implementation of health related social needs (HRSN) screening (e.g., different clinic workflow or staff, different screening triggers, different tools), so that heterogeneity within NCORP practices can be captured
* Clinics must be willing to allow Practice Staff participants to observe the clinical operations in-person

PRACTICE STAFF:

* Must be willing and able to take time to observe in person and document 1-3 selected clinics within the practice (approximately 2-3 hours per clinic)
* Must be staff at the selected and enrolled practice. Suggestions of appropriate staff are cancer care delivery research (CCDR) Lead, research nurse, clinical research coordinator or NCORP Administrators. Staff members with primary clinical roles may also be appropriate, if available
* Must be willing and able to participate in two 1.5 hour virtual training sessions
* Must be willing to interview Clinic Key Informants (approximately 30 minutes per interview; in-person or remotely over the internet or by phone)
* If the clinic is chosen for Part 2, must be willing to schedule an interview between Clinic Key Informant and Wake Forest health HRSN Study Team or designee
* If the clinic is chosen for Part 3, must be willing to participate in a three hour or two 1.5 hour in-person (if possible) workshop(s). If the clinic schedules an in-person workshop, there will be no hybrid or separate virtual option for those that cannot attend
* Must be willing to be recorded when participating in interviews and the workshop.

CLINIC KEY INFORMANT:

* Must be willing to participate in Part 1 Operational Assessment, which involves a semi-structured interview (approximately 30 minutes; in-person or remotely over the internet or by phone) and a brief Non-patient Demographics Survey (approximately 5 minutes)
* If the clinic is chosen for Part 2, must be willing to participate in an additional 45 minute interview (remotely over the internet or by phone)
* If the clinic is chosen for Part 3, must be willing to participate in a three hour or two 1.5 hour in-person (if possible) workshop(s). If the clinic schedules an in-person workshop, there will be no hybrid or separate virtual option for those that cannot attend

Part 3

STAFF WORKSHOP PARTICIPANT:

* Must be a clinic stakeholder (e.g., providers, practice managers, etc.) of the selected clinic
* Must be willing and able to participate in a three hour or two 1.5 hour in-person (if possible) recorded workshop. If the clinic schedules an in-person workshop, there will be no hybrid or separate virtual option for those that cannot attend
* Must be willing to be recorded when participating in interviews and the workshop.

PATIENT WORKSHOP PARTICIPANT:

* Must be a prospective clinic stakeholder (e.g., patient representative) of the selected clinic
* Must be willing and able to participate in a three hour or two 1.5 hour in-person (if possible) recorded workshop. If the clinic schedules an in-person workshop, there will be no hybrid or separate virtual option for those that cannot attend
* Must have received cancer treatment at the selected clinic within the last five years
* Must be willing to be recorded when participating in the workshop.

Exclusion Criteria:

Part 1

PRACTICE STAFF:

** Unable to understand, read and communicate in English, as the trainings and observations will be documented in English

Part 3

STAFF WORKSHOP PARTICIPANT:

** Unable to understand, read and communicate in English, as the workshop will be conducted in English

PATIENT WORKSHOP PARTICIPANT:

** Unable to understand, read and communicate in English, as the workshop will be conducted in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NCI Community Oncology Research Program (NCORP) clinics
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
HRSN screening reach (Part 1) | From study enrollment to approximately 4 and 16 weeks post initial study training
  Determining the perception of the proportion of patients at clinics who are screened for health related social needs (HRSN).
Barriers and facilitators influencing HRSN screening implementation | From study enrollment to time completion of key informant interviews, approximately within 6 months
  Synthesize themes to create a list of barriers and facilitators influencing HRSN screening implementation within high-implementation clinics, moderate-implementation clinics, and low-implementation clinics.
Generation of a tailored implementation plan for each participating clinic | Between time of clinic selection and co-design workshop completion, to be no more than 6 months
  Generation (defined for each clinic as completed or not completed) of a tailored implementation plan for each participating clinic in Part 3 that includes (1) adaptations to current HRSN screening and follow-up processes, and (2) potential implementation strategies to enhance HRSN screening implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, Study Chair — Wake Forest University Health Sciences
Locations (37):
- United States (33):
  - Helen F Graham Cancer Center, Newark, Delaware
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - University Medical Center New Orleans, New Orleans, Louisiana
  - MaineHealth Cancer Care - Brunswick, Brunswick, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Wake Forest NCORP Research Base, Winston-Salem, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- FHP Health Center-Guam, Tamuning, GU, Guam
- Puerto Rico (3):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Wake Forest NCORP Research Base is committed to following the NIH Statement on Sharing Research Data (http://grants.nih.gov/grants/guide/notice-files/NOT-OD-03-032.html). As of July 2018, the WF NCORP RB signed an agreement with NCI to contribute de-identified data and data dictionaries from clinical trials conducted through our RB to the NCI NCTN/NCORP data archive within 6 months of primary and non-primary publications of phase II/III and phase III trials to https://nctn-data-archive.nci.nih.gov/. This will become the primary means for sharing raw data, and we will adhere to the guidelines spelled out in the NCTN/NCORP Data Archive Usage Guide. De-identified data from studies not covered by the agreement (e.g., phase II and observational studies) will be made available upon request. All data files will be de-identified. De-identification procedures will meet the HIPAA criteria as detailed in the Code of Federal Regulations, Part 45, Section 164.514.
Time Frame: 6 months after publication for a 2 year duration
Access Criteria: upon request to NCORP@wakehealth.edu
URL: http://nctn-data-archive.nci.nih.gov/